CLINICAL TRIAL: NCT01209416
Title: The Effect of Pharmacological Antilipolysis on the Metabolic Effects of Ghrelin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: M-2010-0157
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-05

CONDITIONS: Metabolism; Insulin Resistance; Hypopituitarism
Keywords: ghrelin; metabolism; type 2 diabetes; insulin resistance
MeSH Terms: conditions — Insulin Resistance; Hypopituitarism; Diabetes Mellitus, Type 2 | interventions — acipimox; Ghrelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ghrelin / Acipimox (Active Comparator): Ghrelin infusion and tablet acipimox
  Interventions: Drug: Acipimox; Drug: Ghrelin
- Ghrelin / placebo (Active Comparator): Ghrelin infusion and placebo tablets
  Interventions: Drug: Ghrelin; Other: Placebo
- Placebo / Acipimox (Active Comparator): saline infusion and tablet Acipimox
  Interventions: Drug: Acipimox; Other: Placebo
- Placebo / placebo (Placebo Comparator): saline infusion and placebo tablets
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Acipimox — Tablet Acipimox 250 mg administered 4 times previous to and during the investigation day
  Other Names: Tablet Olbetam 250 mg
  Arms: Ghrelin / Acipimox; Placebo / Acipimox
Drug: Ghrelin — Ghrelin infusion 4.2 ng/kg/min throughout the investigation day
  Arms: Ghrelin / Acipimox; Ghrelin / placebo
Other: Placebo — placebo tablets or saline infusion
  Other Names: Placebo tablets; Saline infusion
  Arms: Ghrelin / placebo; Placebo / Acipimox; Placebo / placebo

SUMMARY:
This study will investigate the non-growth-hormone-dependent metabolic effects of the hormone Ghrelin in growth hormone deficient subjects by examining the insulin tolerance as well as signal proteins in fat and muscle biopsies.

DETAILED DESCRIPTION:
Ghrelin is a relatively 'new' hormone that is produced in the stomach and to a lesser extend in the hypothalamus of the brain. The actions of ghrelin are diverse and includes stimulation of the appetite center of the brain and the release of growth hormone. We have for the first time shown that ghrelin also stimulates the metabolism of fatty acids and induces insulin resistance in skeletal muscle. These effects have we confirmed in growth hormone deficient subjects on a stabile substitution treatment with growth hormone and hydrocortisone. With these subjects we can investigate the effects of ghrelin that are independent of growth hormone. The present study is a continuation of these findings, as we wish to investigate whether the insulin resistance effect of ghrelin is dependent of the concomitant metabolism of fatty acids. This is possible by administration of the niacin acid antagonist Acipimox, that blocks the fatty acid metabolism reversibly. We have applied this experimental principle in other settings with success.

Knowledge of the effects of ghrelin in general can in shot-sight as well as in long-sight have great importance for the understanding of growth disorders from overweight and type 2 diabetes to malnutrition and eating disorders.

ELIGIBILITY:
Inclusion Criteria:

* males with hypopituitarism in regard to growth hormone and ACTH in stabile treatment regime
* age 18-65
* BMI 20-35

Exclusion Criteria:

* abuse of alcohol
* malign disease
* medication other than that expected for hypopituitarism
* known disease other than hypopituitarism
* participation in isotope investigations the last 6 months

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2012-06 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Effects of ghrelin during basal and hyperinsulinemic conditions | 5 hours investigation day
  Growth hormone deficient patient investigated with ghrelin infusion and pharmacological antilipolysis (Acipimox) in a randomized cross-over study with 4 study days. During each visit signal proteins in muscle and fat biopsies are investigated with PCR, wester blot and activity assays for ghrelin, growth hormone and insulin. Further is glucose metabolism investigated in basal conditions and during hyperinsulinemic euglycemic clamp.
Effects of ghrelin during basal and hyperinsulinemic conditions | 5 hours investigation day
  Effects of ghrelin on heart rate variability
Effects of ghrelin during basal and hyperinsulinemic conditions | 5 hours investigation day
  Effects of ghrelin on thirst, fluid intake, urine production and natriuresis

CONTACTS AND LOCATIONS:
Overall Officials: Jens Otto L Jørgensen, Professor, Principal Investigator — University Hospital of Aarhus
Locations (1):
- University Hospital of Aarhus, Aarhus, Denmark

REFERENCES:
- [Derived] Jepsen SL, Vestergaard ET, Larraufie P, Gribble FM, Reimann F, Jorgensen JOL, Holst JJ, Kuhre RE. Ghrelin Does Not Directly Stimulate Secretion of Glucagon-like Peptide-1. J Clin Endocrinol Metab. 2020 Jan 1;105(1):266-75. doi: 10.1210/clinem/dgz046. PMID 31608930
- [Derived] Vestergaard ET, Cichosz SL, Moller N, Jorgensen JOL, Fleischer J. Short-term acipimox treatment is associated with decreased cardiac parasympathetic modulation. Br J Clin Pharmacol. 2017 Dec;83(12):2671-2677. doi: 10.1111/bcp.13384. Epub 2017 Aug 24. PMID 28736944
- See also: Original publication on the results from the study — https://www.nature.com/articles/srep42706